CLINICAL TRIAL: NCT06647628
Title: A Randomized, Double Blind Clinical Trial to Assess Safety, Tolerability and Pharmacokinetics of MK-1708 in Healthy Elderly Participants
Brief Title: A Clinical Study of MK-1708 in Healthy Elderly Participants (MK-1708-005)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1708-005
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: 8 participants will be randomized to receive either placebo or MK-1708 dose level 1, then 8 participants will be randomized to receive either placebo or MK-1708 dose level 2.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MK-1708 Dosage 1 (Experimental): Participants receive multiple doses of MK-1708 dosage 1.
  Interventions: Drug: MK-1708
- MK-1708 Dosage 2 (Experimental): Participants receive multiple doses of MK-1708 dosage 2.
  Interventions: Drug: MK-1708
- Placebo (Placebo Comparator): Participants receive multiple doses of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-1708 — MK-1708 oral suspension
  Arms: MK-1708 Dosage 1; MK-1708 Dosage 2
Drug: Placebo — Placebo oral suspension
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn about the safety of MK-1708, and how well elderly people tolerate it. The study will also measure what happens to MK-1708 in a healthy elderly person's body over time (pharmacokinetic or PK study). Researchers will learn if at least 1 dose level of MK-1708 will be safe, well-tolerated, and will be above a certain level in people's blood after 24 hours.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Has a body mass index (BMI) ≥18 and ≤32 kg/m^2, inclusive

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer (malignancy). Participants with definitively treated disease who, in the opinion of the study investigator, are highly unlikely to have a recurrence for the duration of the study may be enrolled at the discretion of the investigator

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with ≥1 adverse event (AE) | Up to 14 days after the last dose
Number of participants discontinuing study therapy due to AE | Up to ~2 weeks
Area under the plasma concentration-time curve from dosing to 24 hours postdose (AUC0-24) of multiple MK-1708 doses | At designated time points up to ~2 weeks
Maximum plasma concentration (Cmax) of multiple MK-1708 doses | At designated time points up to ~20 days
Time to maximum plasma concentration (Tmax) of multiple MK-1708 doses | At designated time points up to ~20 days
Concentration 24 hours postdose (C24) of multiple MK-1708 doses | At designated time points up to ~2 weeks
Apparent oral clearance (CL/F) of multiple MK-1708 doses, at steady state | At designated time points up to ~20 days
Apparent volume of distribution (Vz/F) of multiple MK-1708 doses, at steady state | At designated time points up to ~20 days
Apparent terminal half-life (t½) of multiple MK-1708 doses | At designated time points up to ~20 days
AUC0-24 accumulation ratio of multiple MK-1708 doses | At designated time points up to ~2 weeks
Cmax accumulation ratio of multiple MK-1708 doses | At designated time points up to ~20 days
C24 accumulation ratio of multiple MK-1708 doses | At designated time points up to ~2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Velocity Clinical Research, Hallandale Beach ( Site 0001), Hallandale, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com